CLINICAL TRIAL: NCT06310538
Title: Clinical Study on the Treatment of Breast Hyperplasia With Kou Sha Therapy Based on
Brief Title: Clinical Study on the Treatment of Breast Hyperplasia With Kou Sha Therapy Based on Real World
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hongguo Rong (Other)
Responsible Party: Sponsor-Investigator, Hongguo Rong, Investigator, Beijing University of Chinese Medicine
Organization: Beijing University of Chinese Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024BZYLL0110
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Breast Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kou Sha group (Experimental): Generally, the Kou Sha therapy group needs to kou sha 2-3 times, and after each kou sha, it is necessary to rest for 1 week or all the shas in the part fade before they can be kou sha again. The duration of treatment is 1 menstrual cycle.
  Interventions: Behavioral: kou sha
- Control group (Active Comparator): The control group is treated with conventional Western medicine, and according to the patient's condition, Chinese patent medicine treatment, psychological counseling and lifestyle adjustment are carried out. The duration of treatment is 1 menstrual cycle. Stop all medications during menstruation. During this period, avoid excessive fatigue and mental stimulation, and avoid spicy and irritating foods
  Interventions: Drug: Hongjin Xiaojie Capsules

INTERVENTIONS:
Behavioral: kou sha — Kou sha is one of the most important external treatments in traditional Chinese medicine. By using the kou sha to pat on specific parts of the body or acupuncture points, light or heavy slapping is carried out to produce strong vibrations to relax the meridian qi, promote local blood circulation, and achieve the effect of blood circulation and blood stasis, detoxification and evil spirits.
  Arms: Kou Sha group
Drug: Hongjin Xiaojie Capsules — The main group of HongjinXiaojie capsule is divided into anisanglian, Bupleurum, Notoginseng, golden buckwheat, Xiangfu, chicken Yanteng, etc., which has the effect of soft and hard dispersing knot, soothing liver and regulating Qi, promoting blood circulation and removing blood stasis, reducing swelling and relieving pain, and has a certain effect on the treatment of mammary hyperplasia
  Arms: Control group

SUMMARY:
In this study, epidemiological prospective real-world cohort study design was adopted. The Third Affiliated Hospital of Beijing University of Chinese Medicine and the First Hospital of Handan City, Hebei Province were selected. From the same time appointed before the study, all breast hyperplasia participants who met the admission criteria choosing Kou Sha therapy or routine treatment of western medicine were selected in the sample hospitals.The first 30 participants were included in the planned Kou Sha therapy group while the first 30 participants were included in the control group.Taking the change of the total score of breast pain (McGill Pain Questionnaire Short Form score+breast pain score) as the main curative effect index, and taking McGill pain questionnaire score, breast color ultrasound score, palpation lump score, quality of life, anxiety and depression symptoms, sleep and so on as the secondary curative effect indexes to observe the clinical effect of the method of Kou Sha therapy on breast hyperplasia. The research period is from March 2024 to May 2024.

DETAILED DESCRIPTION:
Investigators adopte a real-world prospective cohort study design to investigate the efficacy and safety of the Kou Sha therapy in the treatment of breast hyperplasia.Kou sha on the key points of breast diseases can dredge the mammary veins, and scraping on the back of the liver, gall bladder, spleen, and stomach can loosen the liver and diarrhea, dredge the internal organs and meridians, regulate emotions, and facilitate the recovery of breast hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of breast hyperplasia, and the course of disease is more than 3 months;
* Female, aged between 18 and 50, with regular menstrual cycle and period, with menstrual cycle of (28±7) d;
* Mild and moderate breast pain, with BI-RADS grade below 4;
* Informed consent, voluntary subjects and signed informed consent.

Exclusion Criteria:

With one of the following circumstances cannot be included in this experimental study:

* Patients with breast malignant tumor, inflammatory disease and other breast diseases;
* Patients with serious primary diseases such as cardiovascular and cerebrovascular diseases, liver, kidney and hematopoietic system are psychotics;
* prepare for women during pregnancy, pregnancy, lactation, menopause, severe menstrual cycle disorder or functional uterine bleeding;
* Severe diabetes, skin trauma or obvious inflammation, redness and ulceration of the skin;
* Diseases with severe bleeding tendency, such as thrombocytopenia, leukemia and allergic purpura;
* Those who are using Chinese and western medicines (including topical medicines, acupuncture, etc.) for the treatment of breast hyperplasia within one month before this treatment or now, and have not used hormonal drugs within half a year;
* Participants in other clinical trials within 3 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Breast pain score | 1 month
  ①Pain score: 0 points for no breast pain, 2 points for mild breast pain, no feeling when not deliberately felt, and no work and life are affected, 4 points for frequent but frequent breast pain that can be tolerated, and slightly affected work and life are counted as 4 points, and obvious persistent breast pain that is unbearable and difficult to work and life to carry out normally is counted as 6 points.
  ②Tender pain score: 0 points for no tenderness, 3 points for slight discomfort after touching and pain after repressing, 6 points for moderate tenderness after touching and aggravation of pain after repressing, obvious pain after touching and pain after slight pressing, and 9 points for unconsciously avoiding pain due to pain when the doctor examines the body.
  The higher the score, the worse the result.
Short Form McGill Pain Inquiry Scale (SF-MPQ) | 1 month
  The higher the score, the worse the result.The scale is divided into 3 parts: ①The pain grading index (PRI) includes 11 sensory words and 4 emotional words, and the degree is divided into 4 levels: none, mild, moderate and severe, with 0, 1, 2 and 3 points, including feeling score (0~36 points) and emotional score (0~9 points), and the PRI sensory score, emotional score and total score can be calculated. ②The visual analogy grading method (VAS) is a 10 cm long straight line, with the two ends representing no pain (0 points) and severe pain (10 points) respectively, in which the patient marks the degree of pain. ③The existing pain intensity (PPI) is divided into 6 grades: no pain, mild discomfort, discomfort, uncomfortable, terrible pain, and extreme pain, with a score of 0, 1, 2, 3, 4, and 5, respectively.

SECONDARY OUTCOMES:
Breast color ultrasound score | 1 month
  The higher the score, the worse the result.Before and after treatment, color ultrasound is used to detect the thickness and echo of the breast gland, the nature and number of breast lumps, the maximum diameter of the breast lump and whether there is a blood flow signal, the number of breast duct dilation, and the number of lymph nodes with enlarged axillary lymph nodes, and the total score is calculated
Palpation lump score | 1 month
  The higher the score, the worse the result.The sum of the lump texture score, the lump distribution range score and the lump size score.
  1. Texture of the lump: 0 points for not touching the obvious thickened lump, 2 points for a small number of palpable hypertrophic glands, slightly tougher for the texture, 4 points for palpable patchy thickened glands, as tough as the tip of the nose, and 6 points for palpable large thickened hard glands, as hard as touching the forehead;
  2. Lump distribution range: 1 point for not palpating local thickened glands in any quadrant of the breast, 2 points for palpating in 1 or 2 quadrants, 4 points for palpating in 3 or 4 quadrants, and 6 points for palpating in 5 or more quadrants.
  3. The size of the lump: 0 points for the local thickened glands or lumps that do not touch the breast, 2 points for the maximum diameter of ≤2 cm, 4 points for the maximum diameter of 2~4 cm, and 6 points for the maximum diameter of >4cm.
Depression symptoms | 1 month
  The higher the score, the worse the result.The Depression Self-Rating Scale (SDS) was used to assess the emotional state of the tester, and a four-level scoring method was used, with higher scores indicating more severe anxiety and depression. The total score is 80 points, which is converted into a 100-point standard score, and the sum of the standard scores of the two scales is calculated.
Anxiety symptoms | 1 month
  The higher the score, the worse the result.The Anxiety Self-Rating Scale (SAS) was used to assess the emotional state of the tester, and a four-level scoring method was used, with higher scores indicating more severe anxiety and depression. The total score is 80 points, which is converted into a 100-point standard score, and the sum of the standard scores of the two scales is calculated.
The quality of life rating scale (QOL) | 1 month
  The quality of life rating scale (QOL) is used for evaluation, which included four dimensions, including physical symptoms, mental health, physical environment, and social function, and each dimension was converted into a standard score of 0~100 points, and the higher the score, the higher the quality of life of the patient.

IPD SHARING:
Plan to Share IPD: No